CLINICAL TRIAL: NCT00652873
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Cabergoline 0.5 mg Tablets and Dostinex 0.5 mg Tablets Administered as 2 x 0.5 mg Tablets in Healthy Adult Females and Males Under Fed Conditions
Brief Title: Bioequivalence Study of Cabergoline Tablets and Dostinex Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Alfred Elvin/Director of biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01211
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: Bioequivalence; Cabergoline; Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received the test product, Cabergoline 0.5 mg tablets under fed conditions
  Interventions: Drug: Cabergoline
- B (Active Comparator): Subjects received the reference product, Dostinex under fed conditions
  Interventions: Drug: Dostinex

INTERVENTIONS:
Drug: Cabergoline — Tablets 0.5 mg (2 x 0.5 mg dose), fed
  Other Names: Dostinex
  Arms: A
Drug: Dostinex — Tablets, 0.5 mg (2 X 0.5 mg dose), fed
  Other Names: Cabergoline
  Arms: B

SUMMARY:
To compare the rate and extent of absorption of cabergoline 0.5 mg tablets (test) versus Dostinex (reference)

DETAILED DESCRIPTION:
To compare the rate and extent of absorption of cabergoline 0.5 mg tablets (test) versus Dostinex (reference) administered as 2 x 0.5 mg tablets under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females or males, smokers or non-smokers
* 18 years of age and older
* Subjects should read, sign and date an Informed Consent Form prior to any study procedures
* Subjects must complete all screening procedures within 28 days prior to the administration of the study medication

Exclusion Criteria:

* Breast feeding female subjects
* Clinically significant anormalities found during medical screening
* Any clinically significant gastrointestinal pathology or unresolved gastrointestinal symptoms susceptible of interfering with the absorption of drugs
* Clinically significant illnesses within 4 weeks of the administration of study medication
* Abnormal laboratory tests judged clinically significant
* ECG abnormalities or vital sign abnormalities at screening
* Subjects with BMI greater than or equal to 30.0
* History of allergic reactions to cabergoline or ergot derivatives
* Any food allergies, intolerances, restrictions, or special diet which in the opinion of the medical subinvestigator, contraindicates the subject's participation in the study
* Positive urine drug screen at screening
* Positive testing for hepatitis B, hepatitis C or HIV at screening
* Positive urine pregnancy test at screening (performed on all females)
* Use of investigational drug or participation in an investigational study, within 30 days prior to administration of the study medication
* Donation of plasma (500 mL) within 7 days or donation or significant loss of whole blood (450 mL) within 56 days prior to the administration of the study medication
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day
* History of drug abuse or use of illegal drugs: use of soft drugs (marijuana, pot) within 3 months of the screening visit or hard drugs (cocaine, PCP, crack)within 1 year of the screening visit
* Subjects who have taken prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption
* Female subjects of childbearing potential who have had unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at last 6 months) within 14 days prior to the study drug administration. The acceptable methods of contraception are condom + spermicide (at least 14 days prior to study drug administration), diaphragm + spermicide (at least 14 days prior to study drug administration)or intrauterine contraceptive device (placed at least 4 weeks prior to study drug administration
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication
* Subjects who have undergone clinically significant surgery within 4 weeks prior to the administration of the study medication
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-07; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 240 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Pharm.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm, Inc., Sainte-Foy, Quebec, Canada